CLINICAL TRIAL: NCT00002231
Title: GENEVAX-HIV (APL 400-003), a Candidate DNA Vaccine: A Pilot Dose Escalation Study of GENEVAX-HIV Delivered Intramuscularly Using the Biojector 2000 in HIV Seronegative Volunteers
Brief Title: Safety and Effects of Giving a New HIV Vaccine (GENEVAX-HIV) to HIV-Negative Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth-Lederle Vaccines (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Prevention
Other Study IDs: 004; 04/400-003-04
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Injections, Intramuscular; HIV Antibodies; Immunity, Cellular; AIDS Vaccines; HIV Seronegativity; Dose-Response Relationship, Immunologic; Vaccines, DNA
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: APL 400-003

SUMMARY:
The purpose of this study is to see if it is safe to give GENEVAX-HIV, a new HIV vaccine, to HIV-negative volunteers. This study will also look at how this vaccine affects the immune system of these volunteers.

DETAILED DESCRIPTION:
In this open-label study, volunteers are given an intramuscular injection of GENEVAX-HIV vaccine using the Biojector 2000. Safety measures and immune response are assessed accordingly.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are 18 - 60 years old.
* Are HIV-negative and in good health.
* Are able to understand how infections such as HIV are spread.
* Agree to use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have hepatitis B or C.
* Have any condition that may prevent you from completing the study.
* Are allergic to bupivacaine, vaccines, or certain local anesthetics.
* Have taken certain medications or have received certain therapies that may affect your immune system.
* Have an immune system disorder or have received therapy for an immune system disorder.
* Have been exposed to HIV within 6 months prior to study entry.
* Have received an experimental HIV vaccine or any other experimental treatment within 30 days prior to study entry.
* Have received blood transfusions within 6 months prior to study entry.
* Abuse alcohol or drugs or have an uncontrolled psychiatric disorder.
* Are pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: RR MacGregor, Study Chair
Locations (1):
- Univ of Pennsylvania Med Ctr, Philadelphia, Pennsylvania, United States